CLINICAL TRIAL: NCT02013427
Title: BRAIN MECHANISMS FOR CLINICAL PLACEBO IN CHRONIC PAIN: A Partially-Blind Randomized Clinical Trial of Placebo and Chronic Back Pain
Brief Title: Placebo In Chronic Back Pain - Double-Blind Randomized Control Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Apkar Apkarian, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00080585; R01AT007987-01A1 (NIH)
Record Dates: First submitted 2013-12-09; First posted 2013-12-17 (Estimated); Results first posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Chronic Low Back Pain
Keywords: chronic; back; pain; brain; MRI
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Pain | interventions — Naproxen; Sugars; Omeprazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Observational (No Intervention): Subjects randomized to this arm will be asked to discontinue their current pain medications for the length of the study. This arm is not blinded, as both study staff and participants will be aware that they are not receiving a study treatment.
- Naproxen & Omeprazole (Active Comparator): Subjects randomized to this arm will be asked to discontinue their current pain medications and take one 500mg naproxen capsule and one 40mg omeprazole capsule twice a day for the length of the study. This arm is double-blind, as neither participants nor study staff will know what medication the participants is receiving (blind to active versus placebo treatment).
  Interventions: Drug: Naproxen; Drug: Omeprazole
- Placebo Only (Placebo Comparator): Subjects randomized to this arm will be asked to discontinue their current pain medications and take two placebo capsules twice a day for the length of the study. This arm is double-blind, as neither participants nor study staff will know what medication the participants is receiving (blind to active versus placebo treatment).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen — Take one 500mg naproxen capsule twice a day.
  Other Names: Aleve; Anaprox; Antalgin; Apranax; Feminax Ultra; Flanax; Inza; Midol Extended Relief; Nalgesin; Naposin; Naprelan; Naprogesic; Naprosyn; Narocin; Proxen; Soproxen; Synflex; Xenobid
  Arms: Naproxen & Omeprazole
Drug: Placebo — Take one placebo capsule twice a day.
  Other Names: Sugar Pill
  Arms: Placebo Only
Drug: Omeprazole — Take one 20mg omeprazole capsule twice a day.
  Other Names: Prilosec; losepine
  Arms: Naproxen & Omeprazole

SUMMARY:
This study is designed to examine brain properties for placebo response in chronic back pain patients. The investigators have preliminary data indicating that, in blinded clinical trial studies with neutral instructions regarding treatment, chronic back pain (CBP) patients can be subdivided into placebo responders and non-responders, and these differences are PREDICTABLE a priori, by brain activity. The results imply that CBP placebo may have clinical utility and that its properties can be studied by human brain imaging techniques. In Phase I of the study, the investigators seek to identify brain imaging parameters that predict the propensity for the placebo response in an independent CBP cohort. In Phase II, the investigators will evaluate the interaction between placebo response and medication treatment in individuals stratified as placebo responders versus non-responders. This research is designed to critically assess the neurobiology of placebo analgesia for chronic pain in a partially-blind clinical trial.

DETAILED DESCRIPTION:
Below is a detailed description of what the study would entail (in other words, what would be expected during each visit for the duration of the study).

* Visit 1 (week -2): Pre-treatment screening (180 min). Participants will complete the informed consent process and are evaluated for inclusion/exclusion criteria. A medical/pain history and physical examination will be completed and participants will be asked to assess current back pain intensity on a VAS scale (0-100mm, no pain to worst possible pain). Participants complete questionnaires and return within 2 weeks for baseline MR imaging scans. Blood will be drawn for a baseline screen to obtain a complete blood count, chemistry panel, and liver function tests. Participants will be asked to discontinue their current pain medications 14 days (2 weeks) prior to their baseline visit and take only acetaminophen rescue medication during this time.
* Visit 2 (week 0): Baseline visit (60-90 min). Participants complete the VAS pain scale, and if their pain is above a designated level and no changes in clinical status are reported, they complete a battery of questionnaires and undergo fMRI procedures (anatomical and functional scans). Participants will then be randomized to one of three groups: active treatment, or placebo, or no-treatment groups; this is done in a partially blind fashion (explained below), with medication dispensed in sufficient quantities until the next visit. The placebo group will receive two placebo capsule bid, and the standard of care group will receive one naproxen capsule (500mg) and one esomeprazole capsule (20 mg) bid for the treatment period. The active and placebo treatment groups are double-blinded, meaning that neither the participant nor the researchers will know which treatment participants are receiving (in part through the use of identical re-encapsulation of study agents). The no-treatment group allocation is not blind, as both participants and study staff will be aware that these participants are not receiving study agent. The no treatment group and all participants assigned to a treatment group will continue to receive rescue medication (n=20).
* Visit 3 (week 2): End of Treatment Period 1/Washout (60-90 min). All procedures will be performed as described for Visit 2. A set of questionnaires will be administered. Adherence will be assessed by pill counts, use of rescue medication documented, and participants will be queried about any side effects experienced. Only rescue medication will be dispensed, to all participants, as they will begin a one week washout of treatment.
* Visit 4 (week 3): End of Washout/Beginning Treatment Period 2 (60-90 min). All procedures will be performed as described for Visit 3, plus the addition of brain scans. Adherence will be assessed by use of rescue medication documented, and participants will be queried about any side effects experienced. Study medication will be dispensed in sufficient quantities until the next visit. All participants remain with the same treatment assignment as in Period 1.
* Visit 5 (week 5): End of Treatment Period 2/Washout 2 (60-90 min). All procedures will be performed as described for Visit 3, with the addition of post-treatment imaging scans. Adherence will be assessed by pill counts, use of rescue medication documented, and participants will be queried about any side effects experienced. Only rescue medication will be dispensed.
* Visit 6 (week 6): End of Washout 2 (90 min). Participants will return to complete questionnaires but no imaging studies will be conducted. Use of rescue medication and side effects will be documented. Exit interviews will be conducted at this time.
* Interim periods: During weeks in between visits, participant data will be tracked with the assistance of a smart phone/computer application designed for the study. Depending upon preference, the research staff will download an app onto participants' phones or give them a link to use on their computers; in the case that a participant does not have a smart phone or easy access to a computer/internet, the study will provide him/her with a smart phone that has the app already installed. Participants will be given a login and will be asked to use this application twice a day right after they take their medication. The app asks participants to rate the severity of their pain and their mood on a Likert scale, and probes them as to whether or not they took their medication.

ELIGIBILITY:
Inclusion Criteria:

* History of low back pain for a minimum of 6 months with signs and symptoms of radiculopathy: positive straight leg raising test with dermatomal radiation and/or myotomal weakness and/or reflex asymmetry; pain must radiate into buttock or below.
* Male or female, age greater than18 years, with no racial/ethnic restrictions.
* Must have a Visual Analog Scale (VAS) pain score >50 mm (of 100 mm maximum) at the baseline visit (for which 0mm = no pain, and 100 mm = worst pain imaginable).
* Must be able to read and speak English and be willing to read and understand instructions as well as questionnaires.
* Must be in generally stable health.
* Must sign an informed consent document after a complete explanation of the study documenting that they understand the purpose of the study, procedures to be undertaken, possible benefits, potential risks, and are willing to participate.

Exclusion Criteria:

* Low back pain associated with any systemic signs or symptoms, e.g., fever, chills.
* Evidence of rheumatoid arthritis, ankylosing spondylitis, acute vertebral fractures, fibromyalgia, history of tumor in the back.
* Other comorbid chronic pain or neurological conditions.
* Involvement in litigation regarding their back pain or having a disability claim or receiving workman's compensation or seeking either as a result of their low back pain.
* Diagnosis of current depression or psychiatric disorder requiring treatment, or such a diagnosis in the previous 6 months.
* Beck Depression Inventory II score of >28.
* Use of therapeutic doses of antidepressant medications (i.e., tricyclic depressants, SSRIs, SNRIs; low doses used for sleep may be allowed).
* Significant other medical disease such as unstable diabetes mellitus, congestive heart failure, coronary or peripheral vascular disease, chronic obstructive lung disease, or malignancy.
* History of gastrointestinal ulcer during the past year.
* History of myocardial infarction in the past year.
* Uncontrolled hypertension.
* Renal insufficiency.
* Allergic to, or non-tolerant of, NSAIDs.
* History of aspirin-sensitive asthma.
* Regular use of low dose aspirin.
* Current use of recreational drugs or history of alcohol or drug abuse.
* Any change in medication for back pain in the last 30 days.
* High dose opioid prophylaxis, as defined as > 50mg morphine equivalent/day.
* Any medical condition that in the investigator's judgment may prevent the individual from completing the study or put the individual at undue risk.
* In the judgment of the investigator, unable or unwilling to follow protocol and instructions.
* Evidence of poor treatment compliance, in the judgment of the investigator.
* Intra-axial implants (e.g. spinal cord stimulators or pumps).
* All exclusion criteria for MR safety: any metallic implants, brain or skull abnormalities, tattoos on large body parts, and claustrophobia.
* Pregnancy, or inability to use an effective form of contraception in women of child-bearing age.
* Diabetes (Type I or Type II).

Prohibited Medications:

* Therapeutic doses of antidepressant medications (i.e., tricyclic depressants, SSRIs, SNRIs; low doses used for sleep may be allowed).
* Oral iron supplementation unless approved by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Apkar Apkarian, PhD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Branco P, Berger S, Abdullah T, Vachon-Presseau E, Cecchi G, Apkarian AV. Predicting placebo analgesia in patients with chronic pain using natural language processing: a preliminary validation study. Pain. 2023 May 1;164(5):1078-1086. doi: 10.1097/j.pain.0000000000002808. Epub 2022 Oct 18. PMID 36524810
- [Derived] Vachon-Presseau E, Abdullah TB, Berger SE, Huang L, Griffith JW, Schnitzer TJ, Apkarian AV. Validating a biosignature-predicting placebo pill response in chronic pain in the settings of a randomized controlled trial. Pain. 2022 May 1;163(5):910-922. doi: 10.1097/j.pain.0000000000002450. PMID 34433773
- [Derived] Berger SE, Branco P, Vachon-Presseau E, Abdullah TB, Cecchi G, Apkarian AV. Quantitative language features identify placebo responders in chronic back pain. Pain. 2021 Jun 1;162(6):1692-1704. doi: 10.1097/j.pain.0000000000002175. PMID 33433145

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observational | Naproxen & Omeprazole | Placebo Only
Started | 25 | 5 | 52
Completed | 20 | 4 | 43
Not Completed | 5 | 1 | 9

BASELINE CHARACTERISTICS:
Population: 25 patients received no treatment. Of the 57 treated individuals, 52 were allocated to placebo treatment (PTx) and 5 were allocated to active treatment (MTX, Naproxen + Esomeprazole) in a double-blind fashion.
  Note: the MTx group was included for blinding purposes (i.e., so that we could tell patients they may receive a placebo or active treatment) hence why the large imbalance between groups. Participants were not informed about the odds for receiving active versus placebo treatment.
Groups:
- Observational- NoTx: Subjects randomized to this arm will be asked to discontinue their current pain medications for the length of the study. This arm is not blinded, as both study staff and participants will be aware that they are not receiving a study treatment.
- PTx (Placebo): Subjects randomized to this arm will be asked to discontinue their current pain medications and take two placebo pills (lactose) capsule twice a day for the length of the study. This arm is double-blind, as neither participants nor study staff will know what medication the participants is receiving (blind to active versus placebo treatment).
  Placebo: Take two placebo capsules twice a day.
- MTx (Naproxen + Omeprazol): Subjects randomized to this arm will be asked to discontinue their current pain medications and take one 500mg naproxen capsule and one 40mg omeprazole capsule twice a day for the length of the study. This arm is double-blind, as neither participants nor study staff will know what medication the participants is receiving (blind to active versus placebo treatment).
  Naproxen: Take one 500mg naproxen capsule twice a day. Omeprazole: Take one 20mg omeprazole capsule twice a day.
- Total: Total of all reporting groups
Arm/Group | Observational- NoTx | PTx (Placebo) | MTx (Naproxen + Omeprazol) | Total
Number analyzed (Participants) | 25 | 52 | 5 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 52 | 5 | 81
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (13.0) | 46.6 (11.7) | 53.8 (5.1) | 47.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 2 | 32
  Male | 13 | 34 | 3 | 50
Region of Enrollment [Number; unit: participants]
  United States | 25 | 52 | 5 | 82

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Assessed by Visual Analogue Scale (VAS)
Description: The primary outcome was changes (% change) in self-reported pain levels using VAS - from 0 (no pain) to 10 (worst imaginable pain).
  Results are presented as largest percentage (%) change in pain before and after the interventions (baseline and post-intervention, 6 weeks).
  Percentage change is calculated with post-intervention pain minus baseline pain, divided by baseline pain i.e. (post - baseline) / baseline.
Time Frame: 6 weeks
Population: 67 patients were randomized into an Observational arm (no treatment, n = 20), Naproxen & Omeprazole (active treatment, n=4) and Placebo only (placebo, n = 43).
Measure: Mean (Standard Deviation); unit: percentage of change in pain
Arm/Group | Observational | Naproxen & Omeprazole | Placebo Only
Number analyzed (Participants) | 20 | 4 | 43
percentage of change in pain | -0.03 (0.14) | -0.10 (0.09) | -0.21 (0.21)

ADVERSE EVENTS:
Time Frame: During the study, the first patient was seen on 11/06/2014, and the last patient was seen on 02/04/2016. The total duration of the study lasted ~15 months. Each participant was in the study for approximately 8 weeks (~56 days).
Description: No serious adverse event (SAE) was reported in the study
Groups:
- PTx (Placebo): Subjects randomized to this arm will be asked to discontinue their current pain medications and take two placebo pills (lactose) twice a day for the length of the study. This arm is double-blind, as neither participants nor study staff will know what medication the participants are receiving (blind to active versus placebo treatment).
  Placebo: Take two placebo capsule twice a day.
- MTx (Naproxen & Omeprazole): Subjects randomized to this arm will be asked to discontinue their current pain medications and take one 500mg naproxen capsule and one 40mg omeprazole capsule twice a day for the length of the study. This arm is double-blind, as neither participants nor study staff will know what medication the participants are receiving (blind to active versus placebo treatment).
  Naproxen: Take one 500mg naproxen capsule twice a day. Omeprazole: Take one 20mg omeprazole capsule twice a day.
Arm/Group | Observational- NoTx | PTx (Placebo) | MTx (Naproxen & Omeprazole)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/52 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/52 | 0/5
Other Adverse Events (participants affected / at risk) | 0/25 | 0/52 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No